CLINICAL TRIAL: NCT01012960
Title: Is the Opioid-induced Pharyngeal and Esophageal Dysfunction Peripherally or Central Mediated?
Brief Title: Opioids and Esophageal Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Johanna Savilampi, MD, Region Örebro County
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: JS001
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Pharyngeal Dysfunction; Esophageal Dysfunction
Keywords: methylnaltrexone; upper esophageal sphincter; lower esophageal sphincter; high resolution solid state manometry; opioid induced pharyngeal and esophageal dysfunction
MeSH Terms: conditions — Esophageal Diseases | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo= normal saline
  Interventions: Drug: methylnaltrexone
- methylnaltexone (Active Comparator): peripheral opioid antagonist
  Interventions: Drug: methylnaltrexone

INTERVENTIONS:
Drug: methylnaltrexone — 0,15 mg/kg sc ( subcutaneously)once per volunteer
  Other Names: Relistor

SUMMARY:
The purpose of this study is to evaluate if opioid-induced effects on the pharynx and esophagus is centrally or peripherally mediated.

DETAILED DESCRIPTION:
Opioids induce pharyngeal and esophageal dysfunction and reduce the lower esophageal sphincter (LES) pressure, and thereby decreases the barrier pressure between the stomach and esophagus. This contributes to an increased risk of regurgitation and aspiration during anaesthesia induction and in the postoperative period, when the patient is treated with opioids for pain relief. The effects of opioid antagonists on the opioid induced pharyngeal dysfunction and lower esophageal sphincter pressure are unknown. Therefore it is of great clinical value to evaluate if these negative effects are reversed by peripheral opioid antagonist, methylnaltrexone.

Methylnaltrexone is one of the newer agents of peripherally acting opioid antagonists that act to reverse some of the side effects of opioid drugs, such as constipation, without affecting analgesia.

If the opioid induced pharyngeal and esophageal dysfunction and reduction of the lower esophageal sphincter pressure is peripherally induced or mediated via peripheral opioid receptors, methylnaltrexone might reverse these effects and thereby reduce postoperative morbidity by reducing pulmonary complications. On the other hand, if the dysfunction is centrally induced and not mediated via peripheral opioid receptors there is no effect of methylnaltrexone.

The pharyngeal and esophageal motility/function can be registered in an easy and objective way with the high resolution manometry, ManoScan 360. ManoScan 360 is an equipment with 36 sensors at 1 cm spacing with 12 tip transducers at every sensor. The 36 closely spaced sensors automatically capture all relevant motor function from the pharynx to the stomach. The system collects reliable and consistent data records with improved diagnostic accuracy, and the data are analyzed using ManoView analyzes software. ManoScan 360 has a CE mark approval and has been used at Örebro University Hospital during the last two years.

ELIGIBILITY:
Inclusion Criteria:

* 18 -40 year old healthy volunteers from both sexes.
* have signed and dated Informed Consent.
* willing and able to comply with the protocol for the duration of the trial.

Exclusion Criteria:

* anamnesis of pharyngoesophageal dysfunction.
* known or history of cardiac, pulmonary or neurological disease.
* ongoing medication.
* allergies to or history of reaction to methylnaltrexone, remifentanil or fentanyl analogues.
* pregnancy or breast feeding.
* participation in another clinical medicinal trial during the last 30 days or where follow-up is not completed.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Does methylnaltrexone influence the upper and lower esophageal sphincter pressure and the swallowing function following opioid administration? | 6 hours per volunteer

SECONDARY OUTCOMES:
Does methylnaltrexone influence the experience of swallowing function following opioid administration? | 6 hours per volunteer

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Wattwil, MD, Principal Investigator — University Hospital Örebro
Locations (2):
- Sweden (2):
  - Department of Anaesthesiology, University Hospital Örebro, Örebro
  - University Hospital Örebro, Örebro

REFERENCES:
- [Derived] Savilampi J, Ahlstrand R, Magnuson A, Wattwil M. Effects of remifentanil on the esophagogastric junction and swallowing. Acta Anaesthesiol Scand. 2013 Sep;57(8):1002-9. doi: 10.1111/aas.12134. Epub 2013 May 29. PMID 23713743